CLINICAL TRIAL: NCT02954003
Title: An Open Label Trial of the Safety and Effectiveness of the ValenTx Endo Bypass System and Use of the Endoscopic Anchor Placement Device in Obese Subjects
Brief Title: The ValenTx Endo Bypass System in Obese Subjects
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: ValenTx, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EN 2.3
Record Dates: First submitted 2016-09-23; First posted 2016-11-03 (Estimated); Last update posted 2016-11-03 (Estimated); Status verified 2016-11

CONDITIONS: Obesity
Keywords: Obesity; Weight Loss
MeSH Terms: conditions — Obesity; Weight Loss

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Endo Bypass (Experimental): Subjects implanted with the investigational ValenTx Endo Bypass System
  Interventions: Device: Endo Bypass System

INTERVENTIONS:
Device: Endo Bypass System — Subject is implanted with the device for up to 3 years.
  Other Names: ValenTx System

SUMMARY:
The purpose of this study is to collect clinical data to support the use of the ValenTx Endo Bypass System to improve weight loss and the resolution of comorbidities in obese subjects.

DETAILED DESCRIPTION:
* Single-arm, non-randomized, open-label, multi-center trial conducted in up to 70 subjects to assess the safety and efficacy of the ValenTx Endo Bypass System over implant duration of up to 36 months.
* Body weight, adverse events and device function in implanted subjects will be monitored at monthly visits for the first year after implant, at quarterly visits during the second year, and biannually during the third year.
* Additional follow-up data will include vital signs, hip and waist circumference, blood lab tests, endoscopic assessments of the condition of the implanted device, and a quality of life questionnaire.
* All subjects will be followed for 12 months after device removal with scheduled visits at 1, 6 and 12 months after explant.
* Subject participation may last up to four years, but is expected to vary with implant duration, which will be determined on a case-by-case basis based on the condition of the implanted device.

ELIGIBILITY:
Inclusion Criteria

1. Between 18- 60 years old.
2. BMI of 40-50 kg/m2 with or without comorbidities, BMI of 35-40 kg/m2 with one or more obesity related comorbidities, or BMI of 30-35 with type 2 diabetes
3. Willing to give informed consent, and able to understand what this means.
4. Documented failure with non-surgical weight loss methods.
5. Willing to follow the study procedures and comply with the visits schedule.
6. Live within a reasonable distance of the research center and be able to attend routine follow up visits.

Exclusion Criteria

1. Pregnancy or intention to become pregnant during the course of the study.
2. Abnormal screening esophagogastroduodenoscopy findings
3. Prior esophageal, gastric or bariatric surgery.
4. Known allergies to any of the device materials.
5. Use of weight loss drugs, stimulants and/or herbal weight loss supplements.
6. Recent or ongoing health conditions that contraindicate undergoing an elective weight loss procedure involving a device implanted within the lumen of the esophagus, stomach and proximal small intestine.
7. Participation in another clinical trial within 60 days of the implant.
8. Presence of psychiatric conditions that would impair the ability to provide informed consent or to comply with study procedures.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2013-12; Primary Completion 2015-10 (Actual); Study Completion 2018-10 (Estimated)

PRIMARY OUTCOMES:
The proportion of subjects affected by serious adverse device effects (SADEs) as defined by International Standards Organization (ISO) standard 14155:2011. | 1 Year
  The proportion of subjects affected by SADEs during the 12 months following their device implant.

SECONDARY OUTCOMES:
Mean 12 Month Weight Loss in Kilograms | 1 Year
  Mean reduction in bodyweight in kilograms from the pre-implant baseline visit to the 12 month post-implant follow-up visit.

CONTACTS AND LOCATIONS:
Overall Officials: Roland Maude-Griffin, Study Director — ValenTx, Inc.
Locations (3):
- Canada (2):
  - St. Joseph Healthcare, Hamilton, Ontario
  - Hopital Laval (IUCPQ), Québec, Quebec
- Hospital San Jose Tec de Monterrey, Monterrey, Nuevo León, Mexico

IPD SHARING:
Plan to Share IPD: No